CLINICAL TRIAL: NCT03290768
Title: Empowering Medicare Patients to Self-Manage Their Type 2 Diabetes Using Continuous Glucose Monitoring (CGM) - Investigational Device Pilot (SMA Investigational Device)
Brief Title: Continuous Glucose Monitors to Regulate Glucose Levels in Type 2 Diabetics - (Protocol 3)
Acronym: CGM_IRB-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Savvysherpa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00022589
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2018-06

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Fitness Trackers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diabetes Management Educational Program (Experimental): Subjects receive a CGM and activity tracker as part of a educational program to help manage their glucose levels.
  Interventions: Device: Continuous Glucose Monitor (CGM); Device: Activity Tracker; Behavioral: Coaching

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — Subjects will use a CGM to develop an understanding of how their behaviors influence their glucose levels.
  Other Names: Dexcom Investigational Use Only (IUO) Device
Device: Activity Tracker — Subjects will use the activity tracker, in combination with a continuous glucose monitor (CGM), to develop an understanding of how their activity levels affect their glucose levels.
  Other Names: Fitbit Charge 2
Behavioral: Coaching — Coaches will help subjects understand the readings from the CGMs and how they are affected by diet choices, use of diabetes medications, etc. Coaches and subjects will have weekly conversations about CGM data and behaviors that affect CGM readings. Coaching will occur via telephone, text messaging, and automated text messaging.

SUMMARY:
This study allows Type 2 diabetics to receive feedback from a continuous glucose monitor (CGM) as part of an educational program designed to help them better manage their glucose levels. Subjects will also wear an activity tracker to monitor their activity and observe its effect on their glucose levels. The educational program will involve calls from coaches to check subjects' progress and answer questions.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with type 2 diabetes
* Be able to read and understand English
* Have access to a telephone
* Have a Medicare Advantage health plan through Senior Dimensions

Exclusion Criteria:

* Pregnant
* Blind
* Deaf
* Receiving chemotherapy or radiation to treat cancer (now or in past 6 months)
* Misusing any drugs (including alcohol, painkillers, hallucinogens, or others)
* Critically ill
* Diagnosed with or experiencing:

  * Kidney disease stages 4 and 5
  * End stage renal disease
  * Severe liver disease
  * Dementia
  * Schizophrenia
  * Bipolar disorder
  * Autism
  * An intellectual or learning disability
  * Arrhythmias other than atrial fibrillation
  * Congestive heart failure
* Has had a:

  * Myocardial infarction within the last 6 months
  * Stroke within the last 6 months
  * Stroke that resulted in significant disability (e.g., unable to write clearly or walk)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 358 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Medical Associates, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetes Management Educational Program
Started | 358
Completed | 193
Not Completed | 165

BASELINE CHARACTERISTICS:
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 358
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants lacked age data.
  years
    number analyzed (Participants) | 356
    (all) | 71.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three participants lacked gender data.
  Participants
    number analyzed (Participants) | 355
    Female | 184
    Male | 171
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 358

OUTCOME MEASURES:

1. Primary Outcome: Program Enrollment Rate (%)
Description: (Number of patients who were shipped devices) / (Number of patients invited to enroll) * 100
Time Frame: up to 9 months
Population: Note that the number analyzed is greater than the number of participants (358) because participants are a subset of those who were invited to participate.
Measure: Number; unit: percentage of invitees
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 5896
percentage of invitees | 6.1

2. Primary Outcome: Program Completion Rate (%)
Description: (Number of patients who complete 10 weeks of CGM) / (Number of patients who received devices) * 100
Time Frame: up to 9 months
Population: Unit of measure, below, should read, "percentage of participants completing 10 weeks of CGM," but there is not enough space.
Measure: Number; unit: percentage of participants
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 358
percentage of participants | 54

3. Secondary Outcome: Weekly Average of Estimated Glucose Values (EGV)
Description: (Sum of EGV for a given week) / (Total number of EGV for a given week)
Time Frame: up to 10 weeks
Population: 358 Participants started the study, but participants dropped out as time passed. By week 10, there were only 193 participants remaining who were providing EGV.
Measure: Mean (Standard Deviation); unit: milligrams/deciliter
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 358
milligrams/deciliter
  Week 1 | 153.9 (59.7)
  Week 2: number analyzed (Participants) | 286
  Week 2 | 152.7 (57.9)
  Week 3: number analyzed (Participants) | 275
  Week 3 | 152.3 (57.1)
  Week 4: number analyzed (Participants) | 266
  Week 4 | 152.9 (57.4)
  Week 5: number analyzed (Participants) | 254
  Week 5 | 151.5 (54.2)
  Week 6: number analyzed (Participants) | 242
  Week 6 | 151.1 (52.3)
  Week 7: number analyzed (Participants) | 225
  Week 7 | 149.9 (52.3)
  Week 8: number analyzed (Participants) | 219
  Week 8 | 149.4 (54.1)
  Week 9: number analyzed (Participants) | 210
  Week 9 | 151.0 (55.6)
  Week 10: number analyzed (Participants) | 193
  Week 10 | 149.6 (54.2)

4. Secondary Outcome: Change in Medication Dosage (mg/Day; U/Day)
Description: (dosage of Rx on Day 180) - (dosage of Rx on Day 0)
Time Frame: up to 9 months
Population: After starting the study, administrator realized that it would not be able to obtain medication data from participants. There is no data to report for this measure.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

5. Secondary Outcome: Average Age of Participants Who Start Trial (Yrs)
Description: (Sum of ages of all enrollees) / (Total number of enrollees)
Time Frame: up to 9 months
Population: Two of the 358 participants who started the study lacked age data.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 356
years | 71.4 (7.6)

6. Secondary Outcome: Average Age of Participants Who Complete Trial (Yrs)
Description: (Sum of age of patients who complete) / (Total number who complete)
Time Frame: up to 9 months
Population: One of the 193 participants who completed 10 weeks of CGM use lacked age data.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 192
years | 70.6 (6.5)

7. Secondary Outcome: Texting With Coaches
Description: (Sum of all text messages) / (Total number of participants*days)
Time Frame: up to 9 months
Measure: Number; unit: text messages per participant per day
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 358
text messages per participant per day | 0.003

8. Secondary Outcome: Coaching Participation Rate
Description: (Sum of weekly coaching calls completed) / (Total number of participants*weeks)
Time Frame: up to 9 months
Measure: Number; unit: calls per participant per week
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 358
calls per participant per week | 0.46

ADVERSE EVENTS:
Time Frame: 10 weeks per participant
Arm/Group | Diabetes Management Educational Program
All-Cause Mortality (participants affected / at risk) | 2/358
Serious Adverse Events (participants affected / at risk) | 3/358
Other Adverse Events (participants affected / at risk) | 10/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Management Educational Program (N=358)
Death from Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Death from artherosclerotic and hypertensive heart disease (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Management Educational Program (N=358)
Bleeding at Insertion Site (Injury, poisoning and procedural complications) | 6 (6)
Bruising at Insertion Site (Injury, poisoning and procedural complications) | 2 (2)
Detached/Broken Sensor Wire (Product Issues) | 1 (1)
Redness/Rash at insertion site (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03290768/Prot_SAP_001.pdf